CLINICAL TRIAL: NCT02710474
Title: Family Nurture Intervention in the NICU: A Multi-Site Trial
Brief Title: Family Nurture Intervention in the NICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Einhorn Family Charitable Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AAAQ7504
Record Dates: First submitted 2016-03-07; First posted 2016-03-16 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Premature Birth; Obstetric Labor, Premature
Keywords: preterm birth; NICU; neonatal; kangaroo care; separation stress; family nurture; maternal confidence; maternal competence; calming cycle; infant neurodevelopment; infant psychological development; mother-infant co-regulation; post-partum depression
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature; Depression, Postpartum | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Care (Active Comparator): Preterm infants will receive current Standard Care (SC) in the NICU.
  Interventions: Behavioral: Standard Care
- Intervention (Experimental): Preterm infants will receive Family Nurture Intervention (FNI) in addition to current Standard Care (SC) in the NICU. Specifically, staff will support the parents and facilitate contact between mother and infant during the NICU stay.
  Interventions: Behavioral: Family Nurture Intervention; Behavioral: Standard Care
- Term Controls (Active Comparator): Full term infants will receive current Standard Care (SC) in the NICU. Term Controls (TC)
  Interventions: Behavioral: Standard Care
- Chart Review (Active Comparator): Chart review will be conducted to acquire a comparison group to determine if our study participants differ from the non-study population.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Family Nurture Intervention — Family Nurture Intervention is facilitated by specially trained Nurture Specialists in a randomized controlled trial (RCT) model (Part I) or applied unit-wide (either through dedicated staff or bedside nurses in Part II). Under FNI, specialists or nurses will support the parents and facilitate contact between mother and baby during the infant's NICU stay. The intervention involves calming interactions between mother and infant in the isolette via odor exchange, firm sustained touch and vocal soothing, through calming interactions during holding and feeding via the Calming Cycle and through family sessions designed to engage the help and support of family members for the mother.
  Other Names: FNI
  Arms: Intervention
Behavioral: Standard Care — Established routine care provided on the NICU floor by specially trained health care professionals.
  Other Names: SC

SUMMARY:
The purpose of this study is to compare neurodevelopment and activity in infants born very preterm (26 to 33 6/7 weeks gestational age (GA)) receiving Standard Care (SC) or Family Nurture Intervention (FNI) in the neonatal intensive care unit (NICU).

The study investigator hypothesizes that FNI will improve: i) neonatal electroencephalographic activity ii) maternal caregiving and wellbeing (psychological and physiological), and iii) infant behavior and neurodevelopment at 18 months corrected age (CA).

The study aims to:

- Replicate efficacy from an earlier trial by conducting the study at multiple sites to allow for greater generalizability.

* SC, approximately 90 infants plus the parents
* FNI, approximately 90 infants plus the parents
* Term Controls, approximately 25 infants plus the parents

DETAILED DESCRIPTION:
Increasing number of studies demonstrating the importance of early mother-infant nurturing interaction on long-term outcomes demonstrates the need for a prevention/remedial intervention in the neonatal intensive care unit (NICU). The foremost goal of neonatal intensive care is to ensure survival and medical stability of the infant. Within the NICU, parental involvement in care is necessarily superseded by the healthcare staff's need to assure survival. Thus, a necessary but detrimental separation between mother and infant is created at a critical period when mother-infant connection and synchrony should be developing. The physiological challenges associated with being born too soon, along with disturbances in normal mother-infant interactions, are key factors underlying the risks of premature infants for a broad range of early and midlife disorders.

Not only are preterm infants at increased risk for adverse outcomes (>50%), but up to 40% of mothers of these infants suffer from depression during the postpartum period and many mothers suffer symptoms of trauma and post-traumatic stress. Importantly, fathers of preterm infants are also at increased for postnatal depression. In addition, a recent review of 10 studies found that mothers of preterm infants are at increased risk for subsequent ischemic heart disease, stroke, atherosclerosis, and death due to cardiovascular disease (CVD). Delivery of a preterm infant has long lasting effects on both parents with both mothers and fathers reporting increased parenting stress when their infants reached 7 years of age.

This study will allow examination of the immediate and long-term effects of new approach on the development of preterm infants and cardiovascular risk of their parents.

ELIGIBILITY:
For the FNI and SC Groups (enrolled competitively at across all participating sites)

Inclusion criteria:

* Infant is between 26 and 33 6/7 weeks gestational age upon admission
* Infant is a singleton or twin

Exclusion criteria:

* Infant's attending physician does not recommend enrollment in the study
* Severe congenital anomalies including chromosomal anomalies
* Ultrasound evidence of large parenchymal hemorrhagic infarction (>2 cm, intraventricular hemorrhage grade 3 or 4)
* Infant cardiac anomalies
* Mother has known history of substance abuse, severe psychiatric illness or psychosis
* Status of enrolled subject changes and subject now falls into exclusion criteria
* Mother and/or infant has a medical condition that precludes intervention components
* Mother and/or infant has a contagion that endangers other participants in the study

For the TC Group (enrolled at one site: MSCHONY)

Inclusion Criteria:

* Infant is born between 38-42 weeks gestation
* Infant is singleton or twin

Exclusion criteria:

* Infant's attending physician does not recommend enrollment in the study
* Severe congenital anomalies including chromosomal anomalies
* Ultrasound evidence of large parenchymal hemorrhagic infarction (>2 cm, intraventricular hemorrhage grade 3 or 4)
* Infant cardiac anomalies
* Mother has known history of substance abuse, severe psychiatric illness or psychosis
* Status of enrolled subject changes and subject now falls into exclusion criteria
* Mother and/or infant has a medical condition that precludes intervention components
* Mother and/or infant has a contagion that endangers other participants in the study

Ages: 26 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 461 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
EEG Power in the frontal polar region | Infant Age at 39-41 Weeks gestational age
  Measured in microvolts (µV)^2

SECONDARY OUTCOMES:
EEG Coherence in the left frontal polar to right frontal polar region | Infant Age at 39-41 Weeks gestational age
  Coherence is a number between 0-1, generated by looking at the similarity/differences in activity between brain regions through analysis of electroencephalogram (EEG).
CES-D Score | Up to 18 months
  To examine maternal depression. The Center for Epidemiologic Studies Depression Scale (CES-D) is a 20 item self-report inventory designed to assess current but nonspecific distress rather than clinically diagnosed depression. It is the most frequently used measure in the field of infant research and maternal depression. Items probe for depressive symptoms and attitudes within the past week. The investigators will examine a low-scoring group CES-D = 0, 1, who endorse no distress.
STAI Score | Up to 18 months
  To examine Maternal Anxiety. The State-Trait Anxiety Inventory (STAI) comprises 2 separate self-report scales of 20 items each that measure state and trait anxiety (Spanish version also available). The S-Anxiety Scale (measuring state), has been found to be a sensitive indicator of changes in transitory anxiety experienced by patients in counseling, psychotherapy, and behavior-modification programs, and has been used to assess the level of anxiety induced by unavoidable real-life stressors. The T-Anxiety scale has proven useful for identifying persons who differ in motivation or drive level. The STAI has been used in studies examining parents of hospitalized children, the transition to a maternal role, perception of illness severity in infants, and maternal anxiety during pregnancy and fetal attachment.
Neurobehavioral Assessment of Infants - Bayley Scales of Infant and Toddler Development, Bayley III | 18 Month corrected age Follow-Up
  At the 18 month corrected age follow-up, infants are administered the Bayley Scales of Infant and Toddler Development, Bayley III consisting of three developmental domains: Cognitive, Language (receptive/expressive) and Motor (fine/gross). For each domain, a composite score is provided and is scaled to a mean score of 100 and a standard deviation of 15. A child will receive 1 point for every item successfully completed. The administration of each section will end if the child received 0 points on 5 consecutive items. Scores <70 indicate significant developmental delays and scores <80 indicate mild to moderate developmental delays.
  Cognitive Scale - comprised of 91 items Language Scale - comprised of 97 items Motor Scale - comprised of 138 items

OTHER OUTCOMES:
Welch Emotional Connection Scale | Up to 18 months
  To examine Mother-Infant Emotional Connection. This is a brief, 4-item assessment requiring 5 minutes or less, which assesses the character of the relationship between study mothers and infants. It is filled out by study staff, who rate mothers and infants in a dyadic interaction on their attraction, their motivation to verbally communicate, their sensitivity to each other, their responsivity to each other, and their communication with physical/facial gestures on independent 3-point scales.
Child Behavior Checklist Score | 18 Month corrected age Follow-Up
  The Child Behavior Checklist (CBCL) is a device by which parents rate a child's problem behaviors and competencies. The CBCL can also be used to measure a child's change in behavior over time or following a treatment. The CBCL consists of 100 items.
Modified Checklist for Autism in Toddlers (M-CHAT) Score | 18 Month corrected age Follow-Up
  The M-CHAT is a questionnaire validated for screening toddlers to assess risk for autism spectrum disorders (ASD). It is a 23 yes/no item questionnaire administered to the mother which can be scored in less than two minutes. The investigators will administer the M-CHAT during the 18 month follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Martha G Welch, MD, Principal Investigator — CUMC
Locations (2):
- United States (2):
  - Morgan Stanley Children's Hospital of New York (MSCHONY), New York, New York
  - University Texas Health Science Center San Antonio (UTHSCSA), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Helle N, Barkmann C, Bartz-Seel J, Diehl T, Ehrhardt S, Hendel A, Nestoriuc Y, Schulte-Markwort M, von der Wense A, Bindt C. Very low birth-weight as a risk factor for postpartum depression four to six weeks postbirth in mothers and fathers: Cross-sectional results from a controlled multicentre cohort study. J Affect Disord. 2015 Jul 15;180:154-61. doi: 10.1016/j.jad.2015.04.001. Epub 2015 Apr 10. PMID 25911131
- [Background] Robbins CL, Hutchings Y, Dietz PM, Kuklina EV, Callaghan WM. History of preterm birth and subsequent cardiovascular disease: a systematic review. Am J Obstet Gynecol. 2014 Apr;210(4):285-297. doi: 10.1016/j.ajog.2013.09.020. Epub 2013 Sep 18. PMID 24055578
- [Background] Holditch-Davis D, Bartlett TR, Blickman AL, Miles MS. Posttraumatic stress symptoms in mothers of premature infants. J Obstet Gynecol Neonatal Nurs. 2003 Mar-Apr;32(2):161-71. doi: 10.1177/0884217503252035. PMID 12685667
- [Derived] Welch MG, Grieve PG, Stark RI, Isler JR, Ludwig RJ, Hane AA, Gong A, Darilek U, Austin J, Myers MM. Family nurture intervention increases term age forebrain EEG activity: A multicenter replication trial. Clin Neurophysiol. 2022 Jun;138:52-60. doi: 10.1016/j.clinph.2022.02.018. Epub 2022 Mar 5. PMID 35358769